CLINICAL TRIAL: NCT05601349
Title: Effectiveness of a Telehealth-based Strategy to Improve the Implementation of the Clinical Practice Guide for Lower Limb Amputees by Neurovascular Disease and Trauma: Intervention Trial Randomised by Clusters
Brief Title: TeleEducation for Implementing a Clinical Practice Guideline For Amputees
Acronym: TEFICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Rehabilitacion en Salud (Network)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: GrupoRS005
Record Dates: First submitted 2019-12-26; First posted 2022-11-01 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Clinical Practice Guidelines; Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Below Knee (Injury); Lower Limb Amputation Knee; Lower Limb Ischemia; Diabetes Mellitus; Rehabilitation; Prosthesis User
Keywords: lower limb amputation; clinical practice guidelines; implementation strategies; rehabilitation
MeSH Terms: conditions — Wounds and Injuries; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Community based intervention study randomized by clusters. These studies are differentiated by the method of randomisation, in which a group of individuals is randomly assigned to an intervention as a group or cluster rather than as individuals.
Who Masked: Participant, Outcomes Assessor
Masking Description: Each cluster is conformed by one hospital of middle or higher attention level, the individuals in each cluster don´t know the intervention options, and the outcomes assessor either
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Implementation of the Clinical Practice Guideline (Other): In this group, all participants (cluster) have access to the clinical practice guideline that has been sent to the office responsible for implementing the guideline in the hospital. Due to the characteristics of the intervention in the control group it does not work as a placebo or a sham intervention.
  Interventions: Behavioral: Telehealth-based strategy
- Tele-education strategy (Active Comparator): Tele-educational program consisting of a virtual course with recommendations from the CPG of lower limb amputees, with three modules: Perioperative, rehabilitation and prostheses
  Interventions: Behavioral: Telehealth-based strategy

INTERVENTIONS:
Behavioral: Telehealth-based strategy — Teleducation course, based on the CPG recommendations

SUMMARY:
The publication of a Clinical Practice Guideline (CPG) is often not enough for its correct use in the field of health care. There are barriers to the implementation of the CPG recommendations, including those related to the lack of knowledge or skills on the part of health service providers. Strategies have been proposed to improve the implementation of the CPGs through interventions with different levels of effectiveness, such as the use of reminders, informative meetings, sending educational material, audits, among others. Some of these interventions can be carried out through Telehealth strategies, that is, with remote services. The purpose of this study is to evaluate the effectiveness of a Telehealth program to improve the implementation of the Clinical Practice Guideline for diagnosis and preoperative, intraoperative and postoperative treatment of the amputee, the prescription of the prosthesis and comprehensive rehabilitation, through strategies to publicize the recommendations included in the CPG and train doctors, reducing the barriers related to the lack of knowledge of the CPG. For this, two groups of institutions that provide health services in Antioquia will be compared, randomized according to two interventions: the socialization of the recommendations of the CPG for amputees, against a combined strategy of education through a Telehealth platform and the delivery of educational material. Compliance with prioritized recommendations of the CPG will be evaluated, related to surgical techniques, perioperative practices, the prescription of prosthetic components and referral to services that allow the comprehensive rehabilitation of the person with amputation. Additionally, the theoretical knowledge of the doctors of each participating institution before and after the interventions will be evaluated through a written test.

DETAILED DESCRIPTION:
The effectiveness of the educational program based on telehealth tools (TeleEducation: virtual course with recommendations from the CPG of lower limb amputees, at least four modules: Orthopedics, surgery, rehabilitation and prostheses; TeleAssistance: virtual conference between CPG researchers and professional from selected hospitals and delivery of educational material containing the recommendations of the CPG) compared to the usual socialization of the CPG in an informative meeting to the health personnel of the institutions, will be evaluated by means of a generalized estimated equation model (GEE) for dichotomous variables using the binomial distribution and logit as a link function since the outcomes that will be used will be handled with two coded response options 1 = satisfy 0 = does not satisfy and given the design of conglomerates where the measurements would be correlated.

The investigators are expecting to improve the implementation of the CPG be at least 15% higher than compare the intervention group with the control group.

The effectiveness of a telehealth based strategy is expected to improve the Implementation of the Clinical Practice Guide for diagnosis and preoperative treatment, intraoperative and postoperative period of the amputated person, the prescription of the prosthesis and the comprehensive rehabilitation in health institutions in Antioquia, Colombia, be at least 15% higher than compare the intervention group with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Hospital providing medium and high complexity services in Antioquia that are linked or linked to the telehealth network of the University of Antioquia.

  * Patients with lower limb amputation due to traumatic, vascular or diabetes mellitus that are treated in the aforementioned institutions.
  * Health professionals who use CPG for people with amputation.
  * Hospitals, patients and professionals who agree to participate in the project

Exclusion Criteria:

* Patients who were amputated for other causes not included in the target population of the CPG, such as cancer and congenital.

  * Amputee patients under 16 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of patients who received two stages amputation in severe infection | 1 week
  First stage for infection control and second stage for remodeling and definitive closure of the stump
Rate of patients who received perioperative analgesia | 72 hours
  Perioperative epidural analgesia in patients who are going to be amputated from lower limbs to decrease acute pain of the stump and phantom limb in the period
Rate of patients who received prophylactic antibiotics | 2 hours before the incision until 24 hours after the amputation
  Antibiotic use (Cefazolin or Vancomycin in case of allergy to beta-lactams) from 2 hours before the incision until 24 hours after the amputation
Rate of patients who received transfemoral amputation instead of knee disarticulation | 24 hours
  Transfemoral amputation instead of knee disarticulation
Rate of patients who received myodesis | 24 hours
  Myodesis (Suture of the adductor muscles to the bone through transosseous tunnels)
Rate of patients who received immediate postoperative prosthesis | 24 hours
  verify the order of the immediate prosthesis and if it was manufactured
Rate of patients who received a SACH foot | 3 to 6 months
  Adapt a solid ankle cushion heel (SACH) foot for amputations of the lower limbs above or below the knee and a low expected level of activity (K1 or K2)
Rate of patients who received an articulated foot | 3 to 6 months
  adapt an articulated foot or a dynamic response foot in people with greater activity requirements (K3 / K4) or who must use the prosthesis on irregular or inclined surfaces
Rate of patients who received a prosthetic knee for above knee amputees | 3 to 6 months
  Monocentric knee with manual locking or a knee with load brake in the K1 and monocentric or polycentric knee of fluid control in the K2, K3, K4 was prescribed
Rate of patients who received a prosthetic knee for knee disarticulated amputees | 3 to 6 months
  mechanical polycentric knee was prescribed for disarticulation in K1 and polycentric fluid control for K2, K3, K4
Rate of patients who received occupational therapy | 3 to 6 months
  occupational rehabilitation and ergonomic adaptations
Rate of patients who received comprehensive Rehabilitation | 2 weeks to 12 weeks
  recommends the implementation of a comprehensive rehabilitation process: cardiopulmonary, musculoskeletal, psychosocial, activities of daily living and work

CONTACTS AND LOCATIONS:
Overall Officials: Jesús A Plata Contreras, Principal Investigator — Universidad de Antioquia
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No